CLINICAL TRIAL: NCT04735003
Title: TRans-catheter Interventions for triCuspid Valve Insufficiency: the iTalian Multicentre Study
Brief Title: Transcatheter Interventions for Tricuspid Insufficiency in Italy
Acronym: TRIC-IT
Status: Recruiting | Type: Observational
Sponsor: Marianna Adamo (Other)
Collaborators: San Raffaele University Hospital, Italy (Other)
Responsible Party: Sponsor-Investigator, Marianna Adamo, Principal investigator, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Organization: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Other Study IDs: 581011977013
Record Dates: First submitted 2021-01-16; First posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Tricuspid Valve Insufficiency
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Transcatheter tricuspid valve interventions — Transcatheter repair or replacement to treat tricuspid regurgitation

SUMMARY:
This is an observational, multi-center, retrospective and prospective study collecting data about patients undergoing transcatheter tricuspid valve interventions in a real world clinical environment. The aim is to report clinical characteristics, procedural results and short- and long-term outcomes of patients undergoing transcatheter tricuspid valve interventions in Italian centres.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing transcatheter treatment of tricuspid regurgitation (native valve -with or without previous surgical valve repair - or degenerated bioprosthesis)
2. Patients who are willing and capable of providing informed consent, and participating in all follow-ups associated with this clinical investigation.

Exclusion Criteria:

1. Valve anatomy unsuitable for transcatheter tricuspid valve interventions.
2. Subjects who are unable or not willing to complete follow-up visits and examination for the duration of the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with significant tricuspid regurgitation who need transcatheter tricuspid valve intervention.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-01-30 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
All-cause death | 1-year
Cardiovascular death or heart failure hospitalization | 1-year

SECONDARY OUTCOMES:
Changes in tricuspid regurgitation degree | 30-day, 1-year and 5-year
Changes in NYHA class | 30-day, 1-year and 5-year
Changes in right ventricular dimensions and function | 30-day, 1-year and 5-year
Changes in liver and kidney function | 30-day, 1-year and 5-year
Changes in medical therapy (i.e. diuretic dose) | 30-day, 1-year and 5-year
All-cause death | 30-day
All-cause death | 5-year
Cardiovascular death or heart failure hospitalization | 30-day
Cardiovascular death or heart failure hospitalization | 5-year

CONTACTS AND LOCATIONS:
Locations (1):
- Marianna Adamo, Brescia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No